CLINICAL TRIAL: NCT02728297
Title: Staged Extended Thoracoscopic Sympathicotomy for Palmo-axillo-plantar Hyperhidrosis; a Pilot Study
Brief Title: Staged Extended Thoracoscopic Sympathicotomy for Palmo-axillo-plantar Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mansoura32
Record Dates: First submitted 2016-03-27; First posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Staged ETS (Experimental): Video-assisted endoscopic sympathicotomy from level of T3 to level of T12 on one side
  Interventions: Procedure: Staged ETS

INTERVENTIONS:
Procedure: Staged ETS — Thoracoscopic approach of sympathetic ganglia T3-T12 on one side, retraction of the diaphragm and lung laterally to expose the ganglia then ablation of each ganglion using electrocauterization.

SUMMARY:
Evaluation of staged endoscopic thoracoscopic sympathicotomy in treatment of palmo-axillo-plantar hyperhidrosis

DETAILED DESCRIPTION:
This is a pilot study that investigates the efficacy of video-assisted endoscopic sympathicotomy from the level of T3 to T12 on combined palmar and plantar hyperhidrosis.

Ablation of ascending sympathetic fibers would help alleviating both types of hyperhidrosis in a single setting.

ELIGIBILITY:
Inclusion Criteria:

* patients with combined palmo-axillo-plantar hyperhidrosis of ASA grade I and II

Exclusion Criteria:

* Patients under 16 years.
* Patients with bradycardia (heart rate <80 beats per minute).
* Patients with concomitant lung pathology, frozen mediastinum, pleural effusion, or history of intercostal tube insertion.
* Patients with cardiac problems with ejection fraction less than 60%.
* Patient suffering from isolated palmo-axillary hyperhidrosis not associated with plantar hyperhidrosis.
* Patients suffering from craniofacial hyperhidrosis, either isolated or combined with other areas of hyperhidrosis.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in severity of hyperhidrosis on visual analogue scale at 24 months | 24 months
  decrease in the severity of hyperhidrosis, both palmar and plantar, according to visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D, Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No